CLINICAL TRIAL: NCT06048341
Title: Effects of Sono-guided Femoral Nerve Block in Arthroscopic Surgery for Meniscal Tear Under Spinal Anesthesia: A Randomized Controlled Trial
Brief Title: FNB in Meniscal Tear Under SA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-07-020-001
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Meniscus Tear; Femoral Nerve Block
Keywords: Meniscus Tear; Femoral Nerve Block
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FNB (Experimental): sono-guided femoral nerve injection with 20ml ropivacaine
  Interventions: Procedure: Sono-guided injection; Drug: Ropivacaine injection
- No FNB (Placebo Comparator): sono-guided femoral nerve injection with 20ml 0.9% saline
  Interventions: Procedure: Sono-guided injection; Drug: Saline injection

INTERVENTIONS:
Procedure: Sono-guided injection — After spinal anesthesia, patients will be injected around femoral nerve using ultrasonography.
Drug: Ropivacaine injection — After spinal anesthesia, patients will be injected 20ml ropivacaine around femoral nerve.
  Arms: FNB
Drug: Saline injection — After spinal anesthesia, patients will be injected 20ml 0.9% saline around femoral nerve.
  Arms: No FNB

SUMMARY:
The investigators will compare the results of sono-guided femoral nerve block in arthroscopic surgery for meniscal tear under spinal anesthesia

DETAILED DESCRIPTION:
This study is a randomized controlled trial of 100 patients, who underwent history taking, physical examinations, x-rays, and MRI or ultrasonography, and were diagnosed with meniscal tear from september 2023 to august 2028. The 100 patients will be assigned to Group I (with femoral nerve block) or Group II (without femoral nerve block) under double-blinded randomization. The randomization will be performed by an independent nurse using a computerized random sequence generator. The operators who participated in the procedure will be blinded to the participant's information. Both group will undergo spinal anesthesia for arthroscopic meniscal surgery. After anesthesia, sono-guided femoral nerve block will be performed. The injection for group1 is 20 mL ropivacaine and for groupII is 20 mL 0.9% saline. A visual analog scale (VAS) for pain will be recorded 1, 3, 6, 12, 18, 24, 36, 48 hours after the operation. VAS scores range from 0 to 10, with 0 being no pain and 10 being the most severe pain ever experienced. Injection with ultrasonography will be performed by a single anesthesiologist. 3 orthopedic surgeons will perform the surgery.

ELIGIBILITY:
Inclsuion Criteria:

* individuals who are scheduled to undergo meniscal surgery and must be received sufficient explanation about the research prior to surgery and have provided their informed consent to participate.

Exclusion Criteria:

* who require simultaneous surgery for concomitant cartilage injury, collateral ligament tear.
* who have previously undergone surgical treatment within the knee joint.
* who have declined to participate in the research.
* where medical, surgical, or anesthetic complications occurred during surgery.
* other cases deemed necessary by the researchers.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-18 (Estimated); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
postoperative pain after 24hours | 24hours
  VAS (Visual analog scale) measured 24 hours after operation
  * the unabbreviated scale title: The visual analog scale
  * the minimum and maximum values: 0, 10
  * higher scores mean a worse outcome.

SECONDARY OUTCOMES:
postoperative pain after 1, 3, 6, 12, 18, 48 hours | 1, 3, 6, 12, 18, 48 hours
  VAS (Visual analog scale) score measured 1, 3, 6, 12, 18, 48 hours after operation
  * the unabbreviated scale title: The visual analog scale
  * the minimum and maximum values: 0, 10
  * higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea